CLINICAL TRIAL: NCT01792648
Title: Effects of Almond Intake on Atherogenic Lipoprotein Particles in Individuals With Increased Abdominal Adiposity
Brief Title: Effects of Almond Intake on Atherogenic Lipoprotein Particles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MM2222
Record Dates: First submitted 2012-04-26; First posted 2013-02-15 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Dyslipidemia; Obesity, Abdominal
Keywords: Almond; Carbohydrate; Diet; Cholesterol
MeSH Terms: conditions — Dyslipidemias; Obesity, Abdominal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Reference Diet (Active Comparator)
  Interventions: Other: Standard reference diet
- Almond Supplemented Diet (Experimental)
  Interventions: Other: Almond supplemented diet
- Low Carbohydrate Reference Diet (Active Comparator)
  Interventions: Other: Low carbohydrate reference diet

INTERVENTIONS:
Other: Standard reference diet — 50% energy as carbohydrate, 15% energy as protein, 35% energy as total fat
  Arms: Standard Reference Diet
Other: Almond supplemented diet — 50% energy as carbohydrate, 15% energy as protein, 35% energy as total fat, 20% energy from almonds
  Arms: Almond Supplemented Diet
Other: Low carbohydrate reference diet — 26% energy from carbohydrate, 29% energy from protein, 45% energy from total fat
  Arms: Low Carbohydrate Reference Diet

SUMMARY:
Increased abdominal adiposity is a key feature of metabolic syndrome, which describes a cluster of cardiovascular disease (CVD) risk factors that also includes insulin resistance, high blood pressure and an atherogenic lipoprotein phenotype characterized by increased plasma triglycerides, low HDL-C, and increased levels of small LDL particles. While lifestyle intervention remains the cornerstone for managing obesity and metabolic syndrome, the optimal dietary macronutrient distribution for improving blood lipids and CVD risk remains a topic of controversy. While both low carbohydrate diets and weight reduction are effective for managing atherogenic dyslipidemia, long-term compliance is low, and it becomes imperative to identify alternative dietary approaches.

Increased consumption of almonds has been shown to lower LDL-C, an effect that exceeds that predicted from changes in fatty acid intake. However, although LDL-C lowering by almonds has been demonstrated in patients with diabetes, there have been no trials in non-diabetic patients with abdominal obesity. Moreover, there is limited information of the effects of almond intake on LDL particle subclasses.

The overall objective of the present study is to determine whether lipoprotein measures of CVD risk in individuals with increased abdominal adiposity are reduced by almond supplementation in a diet with overall macronutrient content that conforms to current guidelines. Our main hypothesis is that in these individuals, almond consumption can reduce levels of small and medium LDL particles without the need to restrict dietary carbohydrates to levels below those currently recommended.

This hypothesis will be tested by comparing the lipoprotein effects of an almond-supplemented diet (20%E) with those of two reference diets that do not contain almond products: one with similar content of carbohydrate, protein, and fat (standard reference), and the other in which carbohydrate content is reduced by substitution of protein and monounsaturated fat (low-carbohydrate reference).

We will provide the diets for 3 weeks each in a randomized 3-period crossover design to 40 individuals with increased abdominal adiposity. We will test whether the almond supplemented diet will result in lower levels of lipoprotein measures of CVD risk, specifically LDL-C and small and medium LDL particles, compared to either the standard or low-carbohydrate reference diets.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 or older
* Increased abdominal adiposity as defined by waist circumference ≥102 for men or ≥88 for women.
* Fasting blood sugar (FBS) < 126 mg/dl
* Weight stable for > 3 months.

Exclusion Criteria:

* History of coronary heart disease, cerebrovascular disease, peripheral vascular disease, bleeding disorder, liver or renal disease, diabetes, lung disease, HIV, or cancer (other than skin cancer) in the last 5 years.
* Taking hormones or drugs known to affect lipid metabolism or blood pressure.
* Systolic blood pressure > 160 mm Hg and diastolic blood pressure > 95 mm Hg.
* Body mass index (BMI) > 38 kg/m2
* User of nicotine products or recreational drugs
* Refusal to abstain from alcohol or dietary supplements during the study.
* Total- and LDL-C > 95th percentile for sex and age.
* Fasting triglycerides > 50mg/dl and > 500 mg/dl
* Abnormal thyroid stimulating hormone (TSH) levels.
* Pregnant or breast-feeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Total and LDL cholesterol | 3 weeks, 8 weeks, 13 weeks
  Change in total and LDL cholesterol between each of the 3 test diets
Change in small and medium LDL particles | 3 weeks, 8 weeks, and 13 weeks
  Change in small and medium LDL particles between each of the 3 test diets
Change in apolipoprotein B | 3 weeks, 8 week, 13 weeks
  Change in apolipoprotein B between each of the 3 test diets

SECONDARY OUTCOMES:
Change in total/HDL-cholesterol ratio | 3 weeks, 8 weeks, 13 weeks
  Change in total/HDL-cholesterol ratio between each of the 3 test diets
Change in LDL peak particle diameter | 3 weeks, 8 week, 13 weeks
  Change in LDL peak particle diameter between each of the 3 test diets
Change in plasma triglycerides | 3 weeks, 8 weeks, 13 weeks
  Change in plasma triglycerides between each of the 3 test diets
Change in HDL-cholesterol | 3 weeks, 8 weeks, 13 weeks
  Change in HDL-cholesterol between each of the 3 test diets
Change in large HDL particles | 3 weeks, 8 weeks, 13 weeks
  Change in large HDL particles between each of the 3 test diets
Change in apolipoprotein AI | 3 weeks, 8 weeks, 13 weeks
  Change in apolipoprotein AI between each of the 3 test diets
Change in HOMA-IR | 3 weeks, 8 weeks, 13 weeks
  Change in homeostatic model assessment insulin resistance (HOMA-IR) after each of the 3 test diets

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Krauss, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Cholesterol Research Center, Berkeley, California, United States

REFERENCES:
- [Derived] Williams PT, Bergeron N, Chiu S, Krauss RM. A randomized, controlled trial on the effects of almonds on lipoprotein response to a higher carbohydrate, lower fat diet in men and women with abdominal adiposity. Lipids Health Dis. 2019 Apr 3;18(1):83. doi: 10.1186/s12944-019-1025-4. PMID 30943980